CLINICAL TRIAL: NCT06993220
Title: Multiparametric Assessment of Residual Congestion at Discharge in Patients With Acute Heart Failure
Brief Title: Evaluating Residual Congestion at Discharge in Acute Heart Failure Patients
Status: Recruiting | Type: Observational
Sponsor: Consorci Sanitari Integral (Other)
Responsible Party: Sponsor
Other Study IDs: 24/53
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-05

CONDITIONS: Acute Heart Failure (AHF); Congestive Heart Failure(CHF)
Keywords: acute heart failure; residual congestion; multiparametric assessment; risk stratification
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients hospitalized for acute heart failure
  Interventions: Diagnostic Test: Evaluation of residual congestion at discharge

INTERVENTIONS:
Diagnostic Test: Evaluation of residual congestion at discharge — Evaluation of residual congestion at discharge will be made using:
  * Clinical variables: composite congestion score calculated by summing the individual scores for orthopnoea, jugular venous distension and pedal oedema;
  * Imaging variables: non-invasive left ventricular filling pressure, number of LUS B lines and the presence of pleural effusion, Venous Excess UltraSound (VExUS) score;
  * Laboratory variables: hemoglobin and hematocrit, NT-proBNP, CA-125, ST2, troponin T, creatinine, AST, ALT, Na, K, urea, bilirubin, C-reactive protein.

SUMMARY:
Treatment of congestion is one of the main goals in patients hospitalized for acute heart failure. Nevertheless, current evidence shows that decongestion is often not achieved and that residual congestion at discharge is strongly associated with poor outcomes. While this association has been demonstrated, previous studies have primarily focused on single parameters of congestion (physical examination, biomarkers, or imaging features). The aim of the study is to assess residual congestion at discharge using a multiparametric approach and to compare the prognostic value of each evaluation strategy. Additionally, the analysis will be supported by artificial intelligence to develop a multiparametric prognostic algorithm that can provide an improved predictive model compared to standard statistical approaches.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patients hospitalized for new onset heart failure or worsening heart failure defined by:

  1. Symptoms classified as New York Heart Association class III or IV.
  2. Clinical or instrumental signs of volume overload (e.g., dyspnea with evidence of pulmonary congestion on X-rays or lung ultrasound, pitting edema, and jugular venous distension).
  3. Elevated NT-proBNP levels within the first 24 hours of admission (cutoff values: 450 ng/L for patients < 50 years; >900 ng/L for patients aged 50-75 years; >1800 ng/L for patients >75 years).
* Ability to provide informed consent.

Exclusion Criteria:

* Known diagnosis of septicemia.
* Glomerular filtration rate < 15 ml/min.
* Life expectancy < 6 months.
* Active myocarditis.
* Heart transplant recipients.
* Patients with ventricular assist devices.
* Congenital heart diseases.
* Moderate-to-severe liver disease (Child-Pugh B-C).
* Patients that will not be followed up by the Heart Failure Unit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for acute heart failure
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Worsening heart failure or cardiovascular death | 6 months after hospital discharge
  Occurrence of the composite of cardiovascular death and worsening heart failure (defined as unplanned hospitalization or urgent visit resulting in diuretic intravenous therapy)

SECONDARY OUTCOMES:
all-cause death | 6 months after hospital discharge
time to first heart failure event | 6 months after hospital discharge
number of heart failure events | 6 months after hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Giosafat Spitaleri, M.D., Principal Investigator — Consorci Sanitari Integral
Locations (1):
- Complex Hospitalari Universitari Moisès Broggi, Sant Joan Despí, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No